CLINICAL TRIAL: NCT07196189
Title: Effects of Fecal Microbiota Transplantation From Patients With Eating Disorders on Body Weight Development in Mice
Brief Title: Effects of Fecal Microbiota Transplantation
Acronym: Transmic-TCA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/289/OB; 2020-A02543-36 (Other: ANSM)
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-04

CONDITIONS: Eating Disorders Symptoms
Keywords: intestinal dysbiosis; intestinal physiology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Stool samples used from independent individuals (healthy volunteers or patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients — A clinical examination (weight, height, Body Mass Index calculation) and ED screening using the SCOFF questionnaire will then be carried out, allowing the patients eligibility criteria to be verified. If the patient is included, the self-questionnaire will be completed on site and stool collection will be carried out.
Other: healthy volunteer — A clinical examination (weight, height, Body Mass Index calculation) and ED screening using the SCOFF questionnaire will then be carried out, allowing the volunteer's eligibility criteria to be verified. If the volunteer is included, the self-questionnaire will be completed on site and stool collection will be carried out.

SUMMARY:
The intestinal microbiota plays an essential role in digestion and, through the gut-brain axis, in the regulation of weight gain and eating behavior. The balaEating disorders (EDs) are serious pathologies affecting adolescence and young adults, likely to become chronic, with long-term morbidity and mortality impacts. These pathologies represent a very important public health issue. EDs are defined by the DSM-V classification criteria and include different forms: anorexia nervosa, bulimia nervosa, hyperphagia, and atypical or unspecified forms. The global prevalence of these diseases reaches 8.4% in women and 2.2% in men. These eating disorders lead to numerous psychiatric and somatic complications and have a significant impact on the quality of life and mortality of patients (particularly in anorexic patients). The molecular mechanisms underlying eating disorders are still poorly understood. The etiological origin of these diseases is complex and involves various biological, psychological, and sociocultural factors. The intestinal microbiota, which corresponds to the community of microorganisms living inside the intestine, could be one of these factors. Indeed, the microorganisms of the microbiota interact very closely with intestinal cells but also with distant organs, such as the brain, via nerve communications or the bloodstream. nce and dialogue between the intestinal microbiota and human cells can be altered following changes in the environment, diet, or stress. These disturbances, found among others in patients suffering from eating disorders, can lead to a lasting change in the composition or metabolic activity of the microbiota (dysbiosis), which can have profound repercussions on human physiology. Several clinical studies conducted on patients with anorexia have highlighted the existence of intestinal dysbiosis in these individuals. As with anorexia, the potential role of intestinal dysbiosis in bulimic and binge eating patients remains currently unknown. This dysbiosis could have a harmful effect on intestinal physiology and promote the onset of functional digestive disorders, which are frequently found in patients suffering from eating disorders. This dysbiosis could also lead to a disruption of communication along the gut-brain axis and contribute to the eating disorders observed in these patients.

DETAILED DESCRIPTION:
The hypothesis of this study is that patients suffering from eating disorders exhibit intestinal dysbiosis that impacts intestinal physiology and eating behavior. This project aims to demonstrate the causal link between this dysbiosis and alterations in intestinal physiology and/or behavior by performing intestinal microbiota transplants in mice from patients spanning the entire spectrum of eating disorders (anorexic, bulimic, binge-eating). The onset of functional digestive disorders and eating disorders in these animals will then be assessed. These results will be compared to those obtained after microbiota transplants from healthy individuals.

These fecal microbiota transplant experiments will allow us to demonstrate the potential involvement of the intestinal microbiota in the onset or maintenance of eating disorders and functional digestive disorders associated with eating disorders. The treatment of functional digestive disorders would constitute an interesting strategy to improve the quality of life of patients suffering from ED and increase the effectiveness of current treatments against this class of pathologies. The demonstration of a role of the intestinal microbiota in the onset or maintenance of EDs would open the way to new therapeutic approaches aimed at modulating the intestinal microbiota of patients in order to restore the microorganism/host balance, reduce alterations in intestinal physiology, and restore communication along the gut-brain axis.

ELIGIBILITY:
Inclusion Criteria:

Patients with ED

* Women.
* Aged 18 to 50.
* First consultation in the Nutrition Department of Rouen University Hospital for ED.
* Positive SCOFF with diagnosis of anorexia nervosa, bulimia nervosa, or binge eating disorder.
* Affiliation with a social security plan.
* Patient who has read and understood the information letter and does not object to participating in the study.

Healthy Volunteers

* Women.
* Aged 18 to 50.
* Body mass index between 18.5 and 24.9 kg/m².
* SCOFF test: no positive response.
* No history of ED or active ED (DSM V criteria negative).
* Affiliation with a social security plan.
* Individual who has read and understood the information letter and does not object to participating in the study.

Exclusion Criteria:

Patients with ED

* Men.
* Aged under 18 and over 50.
* Negative SCOFF.
* Patients who have received antibiotic treatment in the last 3 months.
* Patients with a history of IBD or surgical procedures on the digestive tract.
* Patient refuses to participate in the study.
* Persons deprived of liberty by judicial or administrative order.
* Pregnant or breastfeeding women.
* Protected persons (guardianship or curatorship).

Healthy volunteers

* Men.
* Aged under 18 and over 50.
* SCOFF test with at least one positive response.
* History or active ED (DSM V criteria).
* Persons who have received antibiotic treatment in the last 3 months.
* Person with a history of IBD or surgical procedures on the digestive tract.
* Body mass index less than 18.5 or greater than 24.9 kg/m2.
* Pregnant or breastfeeding women.
* Protected persons (guardianship or curatorship).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with eating disorders (ED) first-time consultants in order to limit potential interference from previous medical treatments or nutritional support and healthy volunteers not presenting with eating disorders.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Body weight assessment of mice receiving fecal microbiota from patients suffering from eating disorders | Day 1
  After collecting stool samples from the patient with eating disorders (ED) or the healthy volunteer, a suspension will be created from the stool samples of the patients or healthy volunteers. This suspension will be transplanted by oral gavage into C57Bl/6 mice whose endogenous microbiota will have been previously eliminated by the administration of antibiotics. Over time, the body weight of the transplanted animals will be evaluated. The main objective of this study is to evaluate the evolution of body weight in mice that received a fecal microbiota transplant from patients with eating disorders and to compare it with that of mice that received a microbiota transplant from healthy volunteers.

SECONDARY OUTCOMES:
Evaluating feeding behavior in response to microbiota transplantation from TCA patients in mice | month 1
  Food and water intake will be monitored daily by weighing
Evaluating body composition in response to microbiota transplantation from TCA patients in mice | month 1
  The body composition of the animals will be determined by echo-MRI (determination of fat mass and lean mass).
Evaluating the occurrence of functional digestive disorders in response to microbiota transplantation from TCA patients in mice | month 1
  The occurrence of functional digestive disorders will be assessed by quantifying the efficiency of gastric emptying, the speed of intestinal transit and the water content of feces in grafted mice.
Evaluating feeding behavior in response to microbiota transplantation from healthy volunteer in mice | month 1
  Food and water intake will be monitored daily by weighing
Evaluating body composition in response to microbiota transplantation from healthy volunteer in mice | month 1
  The body composition of the animals will be determined by echo-MRI (determination of fat mass and lean mass).
Evaluating the occurrence of functional digestive disorders in response to microbiota transplantation from healthy volunteer in mice | month 1
  The occurrence of functional digestive disorders will be assessed by quantifying the efficiency of gastric emptying, the speed of intestinal transit and the water content of feces in grafted mice.
To assess the occurrence of anxious/depressive behaviors in response to microbiota transplantation from TCA patients or healthy volunteers | Month 1
  Each parameter measured in mice after microbiota transplantation (body weight, food intake, intestinal transit time, intestinal permeability, behavioral parameters, etc.) will be compared between the different groups of mice (mice receiving a fecal microbiota transplant from a patient suffering from TCA compared to mice receiving a fecal microbiota transplant from healthy volunteers) using one-way or two-way ANOVA tests, with correction for multiple comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.